CLINICAL TRIAL: NCT00994396
Title: Use of Vitamin D to Improve Glucose Metabolism and Reduce Inflammation in Obese Adolescents on a Standard Weight Loss Program
Brief Title: Vitamin D to Improve Glucose Metabolism and Reduce Inflammation in Obese Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1139897
Record Dates: First submitted 2009-10-12; First posted 2009-10-14 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Obesity; Glucose Intolerance; Inflammation
MeSH Terms: conditions — Obesity; Glucose Intolerance; Inflammation | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo pill (Placebo Comparator): Placebo soft gel pills (soy bean oil encapsulated in soft gel comprised of gelatin, glycerin and water) twice per day for 6 mos
  Interventions: Dietary Supplement: Placebo
- Vitamin D (Experimental): 4000 IU vitamin D3 (cholecalciferol) per day for 6 months.
  Interventions: Dietary Supplement: Vitamin D 3 cholecalciferol

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo soft gel pills (soy bean oil encapsulated in soft gel comprised of gelatin, glycerin and water) twice per day for 6 mos.
  Other Names: Reliance Private Label Supplements
  Arms: Placebo pill
Dietary Supplement: Vitamin D 3 cholecalciferol — 4000 IU (2 soft gels at 2000 IU each) vitamin D3 per day for 6 months.
  Other Names: Reliance Private Label Supplements
  Arms: Vitamin D

SUMMARY:
The investigators' project will study the effects of optimizing the vit D status of obese adolescents on markers of glucose metabolism and inflammation.

DETAILED DESCRIPTION:
The alarming rise in pediatric obesity over the past few decades has been associated with an increase in the occurrence of impaired glucose tolerance and inflammation in children and adolescents. These conditions are part of the "metabolic syndrome", and children with risk factors such as these are much more likely to develop cardiovascular disease or diabetes as adults compared with their lean peers. Within the last few years there has been a growing body of evidence that optimizing vitamin D (vit D) status may alleviate these obesity-associated complications. Further, there is also research that shows that the better the vit D status of overweight individuals, the more favorably they respond to dieting by losing more body fat. The prevalence of vit D deficiency/insufficiency in the North American population has been classified as an "epidemic" by experts in the field and obese teens are considered at an even greater risk for deficiency because they tend to store vit D in their fat stores which is not readily mobilized for use by the body. The investigators' project will study the effects of optimizing the vit D status of obese adolescents on markers of glucose metabolism and inflammation. Obese teens attending an established adolescent weight loss clinic will be supplemented with high-dose vit D for 6 months (mos) which will be administered concurrently with their standard medical care and treatment. At baseline, 3 mos and 6 mos the investigators will measure vit D status, serum markers of insulin sensitivity and glucose metabolism; serum markers of inflammation; and body weight/height and waist circumference. At baseline and 6 mos only the investigators also measure body composition (percent body fat by dual-energy x-ray absorptiometry) and confounding lifestyle factors known to affect vit D, glucose metabolism or inflammation (e.g., nutrient intake, physical activity, sun exposure, pubertal stage). Results gleaned from this study will help to advance the prevention and treatment of obesity-related complications and have the potential to lead to significant reductions in healthcare costs and co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Obese adolescent (BMI > 85th percentile for age)
* 9-19 years of age
* attending the ADOBE clinic at the University of Missouri

Exclusion Criteria:

* use of vit D supplements other than standard multi-vitamin preparation
* (i.e., should not be receiving vit D > 1000 IU/d) use of medications that interfere with vit D metabolism (e.g., anti-convulsive)
* history of hepatic or renal disorders;
* undergoing ultraviolet radiation as medical therapy;
* pregnancy;
* cigarette smoking;
* current use of commercial tanning bed;

Ages: 9 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2009-11; Primary Completion 2011-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
serum 25-hydroxy vitamin D concentrations | baseline, 3, 6 months
serum concentrations of inflammatory markers (Interleukin-6, TNF-alpha, c reactive protein) | baseline and 6 mos
Hemoglobin A1C, serum glucose and insulin concentrations | baseline, 3 and 6 months

SECONDARY OUTCOMES:
Body composition as measured by DXA | baseline and 6 mos
Body mass index | baseline, 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine A Peterson, Ph.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Belenchia AM, Tosh AK, Hillman LS, Peterson CA. Correcting vitamin D insufficiency improves insulin sensitivity in obese adolescents: a randomized controlled trial. Am J Clin Nutr. 2013 Apr;97(4):774-81. doi: 10.3945/ajcn.112.050013. Epub 2013 Feb 13. PMID 23407306